CLINICAL TRIAL: NCT01572428
Title: Randomized Controlled Trial Comparing the Use of Narrow-Band Imaging Versus Standard White Light for the Detection of Serrated Lesions in the Proximal Colon
Brief Title: Narrow-Band Imaging Versus Standard White Light for the Detection of Serrated Lesions in the Proximal Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Douglas K. Rex, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1012-17
Record Dates: First submitted 2011-07-11; First posted 2012-04-06 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Colon Cancer
Keywords: Proximal Colon Cancer; Serrated Colon Lesions; Narrow Band Imaging
MeSH Terms: conditions — Colonic Neoplasms | interventions — Watchful Waiting; Narrow Band Imaging; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrow-Band Imaging (NBI) (Active Comparator): Inspection with Narrow-Band Imaging(NBI) versus inspection with standard white light(usual care)
  Interventions: Procedure: Inspection with Narrow-Band Imaging(NBI)
- Standard White Light (Active Comparator): Inspection with Standard White Light versus Narrow-Band Imaging(NBI)
  Interventions: Procedure: Inspection with Narrow-Band Imaging(NBI); Procedure: Standard White Light

INTERVENTIONS:
Procedure: Inspection with Narrow-Band Imaging(NBI) — Narrow-Band Imaging(NBI)of the colon rather than the standard white light in the inspection of the colon during colonoscopy.
  Other Names: Colonoscopy
Procedure: Standard White Light — Use of Standard White Light on the colon rather than Narrow-Band Imaging(NBI)in the inspection of the colon during a colonoscopy.
  Other Names: Colonoscopy
  Arms: Standard White Light

SUMMARY:
This is a study to determine if using Narrow-Band Imaging of the colon, rather than the usual white light on the colon, will improve the detection of a type of polyp called serrated. The polyps are called serrated because of their appearance under the microscope after they have been removed. They tend to be located up high in the colon, far away from the rectum. They have been definitely shown to be a type of precancerous polyp and it is possible that using Narrow-Band Imaging will make it easier to see them, as they can be quite difficult to see with standard white light.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing the use of Narrow-Band Imaging (illumination of the colon in blue light)versus standard white light for the detection of serrated lesions in the proximal colon (the colon proximal to the splenic flexure). Recent studies have indicated that colonoscopy is more effective in preventing cancer in the left side of the colon than the right side of the colon. The reasons for this difference may be partly biologic, in that a special group of polyps known as serrated polyps, particularly sessile serrated adenomas, are located primarily proximal to the splenic flexure. These lesions share molecular features with a group of cancers that occur primarily in the proximal colon. These molecular features include CpG island methylator phenotype (CIMP) and microsatellite instability. These lesions are endoscopically subtle in that they are often flat, have the same color as the surrounding mucosa, and are hard to differentiate from normal mucosa. Narrow-Band Imaging has anecdotally been used to highlight the appearance of these lesions. This study will test whether Narrow-Band Imaging increases the detection of serrated lesions in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-85
* Intact colon and rectum
* American Society of Anesthesiology risk class 1, 2 or 3

Exclusion Criteria:

* No prior surgical resection of colon or rectum

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07-07 (Actual); Study Completion 2014-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Beltway Surgical Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Rex DK, Clodfelter R, Rahmani F, Fatima H, James-Stevenson TN, Tang JC, Kim HN, McHenry L, Kahi CJ, Rogers NA, Helper DJ, Sagi SV, Kessler WR, Wo JM, Fischer M, Kwo PY. Narrow-band imaging versus white light for the detection of proximal colon serrated lesions: a randomized, controlled trial. Gastrointest Endosc. 2016 Jan;83(1):166-71. doi: 10.1016/j.gie.2015.03.1915. Epub 2015 May 5. PMID 25952085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of patients enrolled(898) differs from number of patients started(804). This is because 94 patients were enrolled but not randomized for various reasons such as inadequate bowel preparation, research personnel/scope not being available, ineligibility of patient per colonoscopist discretion, patient withdrawing consent prior to randomization.
Period: Overall Study
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
Started | 402 | 402
Completed | 399 | 401
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light | Total
Number analyzed (Participants) | 399 | 401 | 800
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.08 (8.294) | 61.41 (8.251) | 61.25 (8.269)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 240 | 456
  Male | 183 | 161 | 344
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 339 | 329 | 668
  Black or African American | 54 | 63 | 117
  Other | 4 | 3 | 7
  Unknown | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 399 | 401 | 800
Tobacco use [Count of Participants; unit: Participants]
  Current | 53 | 44 | 97
  Past | 130 | 123 | 253
  Never | 216 | 234 | 450
ASA risk class [Count of Participants; unit: Participants] — ASA 1 -- a normal healthy patient ASA 2 -- a patient with mild systemic disease ASA 3 -- a patient with severe systemic disease
  Participants
    1 | 52 | 63 | 115
    2 | 230 | 226 | 456
    3 | 117 | 112 | 229
Indication [Count of Participants; unit: Participants]
  Screening | 212 | 203 | 415
  Surveillance | 149 | 162 | 311
  Other | 38 | 36 | 74
Time from end of colon prep to procedure start [Mean (Standard Deviation); unit: Hours] | 6.12 (2.41) | 6.10 (1.99) | 6.11 (2.21)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Serrated Lesions Proximal to the Sigmoid Colon
Description: Total quantity of serrated lesions found proximal to the sigmoid colon during colonoscopy.
Time Frame: During the colonoscopy procedure
Measure: Number; unit: Serrated Lesions
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
Number analyzed (Participants) | 399 | 401
Serrated Lesions
  Any size | 204 | 158
  Greater than 5mm in size | 95 | 59
  Greater than or equal to 10mm | 39 | 20

2. Primary Outcome: Number of Serrated Lesions Proximal to the Sigmoid Colon Per Patient
Description: Average number of polyps per patient that had serrated histology and were located proximal to the sigmoid colon (cecum to transverse colon).
Time Frame: During the colonoscopy procedure
Measure: Mean (Standard Deviation); unit: Number of serrated lesions
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
Number analyzed (Participants) | 399 | 401
Number of serrated lesions
  Any size | 0.51 (1.18) | 0.39 (0.76)
  Greater than 5mm in size | 0.24 (0.70) | 0.15 (0.45)
  Greater than or equal to 10mm | 0.10 (0.42) | 0.05 (0.23)

3. Secondary Outcome: Patients With 1 or More Serrated Lesions Proximal to the Sigmoid Colon
Description: Patient had to have at least 1 polyp that had serrated histology and was located proximal to the sigmoid colon (cecum to transverse colon).
Time Frame: During the colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
Number analyzed (Participants) | 399 | 401
Participants
  Any size | 105 | 107
  Greater than 5mm in size | 60 | 45
  Greater than or equal to 10mm | 25 | 19

4. Secondary Outcome: Total Number of Conventional Adenomas in Entire Colon
Description: Total quantity of adenomas found during colonoscopy procedure.
Time Frame: During the colonoscopy procedure
Measure: Number; unit: Conventional Adenomas
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
Number analyzed (Participants) | 399 | 401
Conventional Adenomas
  All Sizes | 438 | 434
  Greater than 5mm in size | 110 | 90
  Greater than or equal to 10mm | 29 | 22

5. Secondary Outcome: Number of Conventional Adenomas Per Patient in Entire Colon
Description: Average number of adenomas (located anywhere throughout the colon) found per patient.
Time Frame: During the colonoscopy procedure
Measure: Mean (Standard Deviation); unit: Adenomas per patient
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
Number analyzed (Participants) | 399 | 401
Adenomas per patient
  All Sizes | 1.1 (1.61) | 1.08 (1.72)
  Greater than 5mm in size | 0.28 (0.62) | 0.22 (0.67)
  Greater than or equal to 10mm | 0.07 (0.30) | 0.05 (0.27)

6. Secondary Outcome: Patients With 1 or More Conventional Adenomas
Description: Patient had to have at least 1 polyp that was an adenoma.
Time Frame: During the colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
Number analyzed (Participants) | 399 | 401
Participants
  Any size | 202 | 189
  Greater than 5mm in size | 84 | 61
  Greater than or equal to 10mm | 25 | 18

ADVERSE EVENTS:
Time Frame: 38 months
Arm/Group | Narrow-Band Imaging (NBI) | Standard White Light
All-Cause Mortality (participants affected / at risk) | 0/399 | 0/401
Serious Adverse Events (participants affected / at risk) | 0/399 | 0/401
Other Adverse Events (participants affected / at risk) | 0/399 | 0/401

LIMITATIONS AND CAVEATS:
Endoscopists weren't blinded to the type of light being used during withdrawal, which is a limitation of all detection studies. Number of SSPs were not specifically an endpoint of the study, but rather the entire serrated class of polyps.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No